CLINICAL TRIAL: NCT00723099
Title: Transplantation of Umbilical Cord Blood in Patients With Hematological Malignancies Using a Reduced-Intensity Preparative Regimen (A Multi-Center Trial Coordinated by the FHCRC)
Brief Title: Donor Umbilical Cord Blood Transplant in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2239.00; NCI-2009-01551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2239 (Other: Fred Hutch/University of Washington Cancer Consortium); 2239.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Aggressive Non-Hodgkin Lymphoma; Chronic Myelogenous Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Indolent Non-Hodgkin Lymphoma; Lymphoma; Mixed Phenotype Acute Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Recurrent Chronic Lymphocytic Leukemia; Recurrent Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Plasma Cell Myeloma; Recurrent Small Lymphocytic Lymphoma; Recurrent T-Cell Non-Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Chronic Myelogenous Leukemia; Refractory Follicular Lymphoma; Refractory Hodgkin Lymphoma; Refractory Lymphoplasmacytic Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Small Lymphocytic Lymphoma; T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Lymphoma; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Multiple Myeloma; Lymphoma, T-Cell; Hodgkin Disease | interventions — Cyclophosphamide; Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, transplant) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6. Patients undergo a lower dose of TBI on day -1.
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.
  IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days 0 to +180 and mycophenolate mofetil IV or PO every 8 hours on days -3 to +96.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo umbilical cord blood transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cyclosporine — Given IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation
Procedure: Umbilical Cord Blood Transplantation — Undergo umbilical cord blood transplant
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This phase II trial is studying how well umbilical cord blood transplant from a donor works in treating patients with hematological cancer. Giving chemotherapy and total-body irradiation (TBI) before a donor umbilical cord blood transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from an unrelated donor, that do not exactly match the patient's blood, are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate probability of one year survival.

II. Demonstrate equivalent or improved engraftment rates with a non-anti-thymocyte globulin (ATG) based conditioning regimen. Patients will be considered graft failure/rejections provided they meet any of the criteria listed below:

* Absence of 3 consecutive days with neutrophils >= 500/ul combined with host cluster of differentiation (CD)3 peripheral blood chimerism >= 50% at day 42
* Absence of 3 consecutive days with neutrophils >= 500/ul under any circumstances at day 55
* Death after day 28 with neutrophil count < 100/ul without any evidence of engraftment (< 5% donor CD3)
* Primary autologous count recovery with < 5% donor CD3 peripheral blood chimerism at count recovery and without relapse

SECONDARY OBJECTIVES:

I. Six month non-relapse mortality.

II. Overall incidence of graft failure/rejection. Patients will be considered graft failure/rejections provided they meet any of the criteria listed below:

* Absence of 3 consecutive days with neutrophils >= 500/ul combined with host CD3 peripheral blood chimerism >= 50% at day 42
* Absence of 3 consecutive days with neutrophils >= 500/ul under any circumstances at day 55
* Death after day 28 with neutrophil count < 100/ul without any evidence of engraftment (< 5% donor CD3)
* Primary autologous count recovery with < 5% donor CD3 peripheral blood chimerism at count recovery and without relapse

III. Kinetics of chimeric reconstitution.

IV. Incidence of neutrophil engraftment by day 42.

V. Incidence of platelet engraftment by six months.

VI. Incidence of grade II-IV and III-IV acute graft-versus-host disease (GvHD) at day 100.

VII. Incidence of one year chronic GvHD.

VIII. Incidence of clinically significant infections at 6 months, 1 year, 2 years.

IX. Probability of one and two year survival.

X. Incidence of one and two year relapse or disease progression.

XI. Fred Hutchinson Cancer Research Center (FHCRC) patients: Kinetics of immune reconstitution, with both functional and quantitative assays.

XII. FHCRC patients: Examination of possible immunologic factors leading to emergence of a dominant unit.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6. Patients undergo a lower dose of total-body irradiation (TBI) on day -1.

UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.

IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days -3 to +180 and mycophenolate mofetil IV or orally (PO) every 8 hours on days 0 to +96.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 70 may be considered if performance status > 80% or Eastern Cooperative Oncology Group (ECOG) =< 1 and comorbidity score < 3; these patients must be discussed with the principal investigator (PI), Rachel Salit prior to enrollment
* Adequate cardiac function defined as absence of decompensated congestive heart failure, or uncontrolled arrhythmia and:

  * Left ventricular ejection fraction >= 35% or
  * Fractional shortening > 22%
* Adequate pulmonary function defined as diffusion capacity of carbon monoxide (DLCO) > 30% predicted, and absence of oxygen (O2) requirements
* Adequate hepatic function; patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, histology, and the degree of portal hypertension; patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* Adequate renal function defined as creatinine =< 2.0 mg/dl (adults) or creatinine clearance > 40 ml/min (pediatrics)
* All adults with a creatinine > 1.2 or a history of renal dysfunction must have estimated creatinine clearance > 40 ml/min
* Performance status score: Karnofsky (for adults) >= 60 or ECOG 0-2; Lansky (for children) score >= 50
* If recent mold infection, e.g., Aspergillus, must be cleared by infectious disease
* Second hematopoietic cell transplant: Must be >= 3 months after prior myeloablative transplant
* Patients who have received < 2 cycles of multiagent chemotherapy and patients who have received no multiagent chemotherapy within the 3 months previous to umbilical cord blood transplant (UCBT) as well as patients experiencing graft failure following previous allogeneic transplant
* Acute myeloid leukemia/acute lymphoblastic leukemia, including biphenotypic acute leukemia or mixed-lineage leukemia: Must have < 5% morphologic marrow blasts in an evaluable marrow (> 25% of normal cellularity for age) collected less than one month prior to start of conditioning; patients persistently aplastic for greater than one month since completing last chemotherapy are also eligible with the approval of the PI or designee
* Chronic myelogenous leukemia: All types, except refractory blast crisis; chronic phase patients must have failed or been intolerant to Gleevec or other tyrosine kinase inhibitors; at time of transplant, patients must have < 5% blasts in an evaluable marrow (> 25% of normal cellularity for age) by morphology within the bone marrow
* Myelodysplastic syndrome (MDS): Any subtype; morphologic blasts must be less than 5% in an evaluable marrow (> 25% of normal cellularity for age); if blasts are 5% or more, patient requires induction chemotherapy pre-transplant to reduce blast count to less than 5%; patients who have a hypocellular marrow in the absence of excess blasts that is related to the underlying disease or as a result of treatment for MDS may also be eligible with the approval of the PI or designee
* Large-cell lymphoma and aggressive T-cell lymphoma: With chemotherapy sensitive disease that has failed autologous transplant or patients who are ineligible for an autologous transplant; chemotherapy sensitive disease is defined as >= 50% reduction in the size of the tumor with the chemotherapy regimen immediately preceding transplant
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL): Must be refractory to fludarabine (fludarabine phosphate) or fail to have a complete or partial response after therapy with a regimen containing fludarabine (or another nucleoside analog, e.g. cladribine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing fludarabine (or another nucleoside analog)
* Hodgkin disease: Must have received and failed frontline therapy
* Follicular lymphoma, marginal zone B-cell lymphoma, lymphoplasmacytic lymphoma, mantle-cell lymphoma, and indolent T-cell lymphomas: Must have progressed with the most recent remission duration being < 6 months; patients with bulky disease should be considered for debulking chemotherapy before transplant; patients with refractory disease are eligible, unless they have bulky disease and an estimated tumor doubling time of less than one month
* Multiple myeloma: Must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative hematopoietic cell transplant (HCT) is permitted
* Myeloproliferative syndromes
* DONOR: Cord blood (CB) donor selection will be based on institutional guidelines and in general should be selected to optimize both human leukocyte antigen (HLA) match and cell dose; additionally, CB grafts shall consist of one or two CB donors based on, but not exclusively determined by, cell dose (total nucleated cell [TNC]/kg and CD34/kg), HLA matching and disease status and indication for transplant; attending preference will be allowed for single versus double unit as well as the degree of mismatching based on patient specific factors, as long as the following minimum criteria are met:

  * HLA matching

    * Minimum requirement: The CB graft(s) must be matched at a minimum at 4/6 HLA-A, B, DRB1 loci with the recipient. Therefore 0-2 mismatches at the A or B or DRB1 loci based on intermediate resolution A, B antigen and DRB1 allele typing for determination of HLA-match is allowed
    * HLA-matching determined by high-resolution typing is allowed per institutional guidelines as long as the minimum criteria are met
  * Selection of two CB units is mandatory when a single cord blood unit does not meet the following criteria:

    * Match grade 6/6; TNC Dose >= 2.5 x 10^7/kg
    * Match grade 5/6 or 4/6; TNC dose >= 4.0 (+/- 0.5) x 10^7/kg
  * If two CB units are used, the total cell dose of the combined units must be at least 3.0 x 10^7 TNC per kilogram recipient weight based on pre-cryopreservation numbers, with each CB unit containing a MINIMUM of 1.5 x 10^7 TNC/kg
  * The minimum recommended CD34/kg cell dose should be 2 x 10^5 CD34/kg, total dose from a single or combined double
  * The unmanipulated CB unit(s) will be Food and Drug Administration (FDA) licensed or will be obtained under a separate investigational new drug (IND), such as the National Marrow Donor Program (NMDP) Protocol 10-CBA conducted under BB IND-7555 or another IND sponsored by (1) a participating institution or (2) an investigator at FHCRC or one of the participating institutions
  * FHCRC only: Up to 5% of cord blood product, when ready for infusion, may be withheld for research purposes as long as thresholds for infused TNC dose are met; threshold for double unit transplantation is >= 3.0 x 10^7/kg; these products will be used to conduct studies involving the immunobiology of double cord transplantation and kinetics of engraftment

Exclusion Criteria:

* Patients with an available 5-6/6 HLA-A, B, DRB1 matched sibling donor
* Pregnancy or breastfeeding
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* Active central nervous system malignancy
* Patients who have received >= 2 cycles of multiagent chemotherapy within the 3 months previous to UCBT; patients who have had previous autologous transplant within 12 months of UCBT are excluded regardless of history of recent treatment
* DONOR: Any cord blood units with < 1.5 x 10^7 total nucleated cells per kilogram recipient weight
* DONOR: Any cord blood units without the full maternal testing and negative results for hepatitis A, B, C, HIV, and human T-lymphotropic virus (HTLV-1) viruses; any additional available virology results on the unit itself will be reviewed but are not mandated, complete or always available; cord blood units are presumed to be cytomegalovirus (CMV) negative regardless of serologic testing due to passive transmission of maternal CMV antibodies

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-06-25 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Salit, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - University of Colorado Hospital, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - LDS Hospital, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 and 2 Treatment: CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6.
  Arm 1 (patients with lower risk of graft failure-have received multi-agent chemotherapy in the prior 2 months or history of prior autologous transplant): Patients undergo 200 cGy TBI on day -1.
  Arm 2 (patients at higher risk of graft failure-have not received multi agent chemotherapy in the prior 2 months and no history of prior autologous transplant): Patients undergo 300 cGy TBI on day -1
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.
  IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days 0 to +180 and mycophenolate mofetil IV or PO every 8 hours on days -3 to +96.
Period: Overall Study
Arm/Group | Arm 1 and 2 Treatment
Started | 73
Completed | 72
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Chemotherapy, Transplant): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6.
  ARM 1(patients at low risk for graft failure) - patients receive 200cGy TBI ARM 2 (patients at high risk for graft failure) - patients receive 300cGy TBI
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.
  IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days 0 to +180 and mycophenolate mofetil IV or PO every 8 hours on days -3 to +96.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo single or double umbilical cord blood transplant
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] — Patients > 70 may be considered if performance status > 80% or Eastern Cooperative Oncology Group (ECOG) =< 1 and comorbidity score < 3; these patients must be discussed with the principal investigator (PI), Rachel Salit prior to enrollment
  years | 60 [13 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 54
  More than one race | 2
  Unknown or Not Reported | 2
Karnofsky Performance Scale [Count of Participants; unit: Participants] — Scale from 0-100 with
  100= Normal no complaints 90= Normal activity with minor signs or symptoms of disease 80= Normal activity with effort, some signs or symptoms of disease 70= Cares for self, unable to carry on normal activity 60= Requires occasional assistance 50= Requires considerable assistance 40= Disabled 30= Severely disabled 20= Very sick, hospitalized 10= Moribund 0= Dead
  Participants
    100 | 17
    90 | 29
    80 | 18
    70 | 6
    50 | 1
    unknown | 1
Hematopoeitic Cell Transplant Comorbidity Index [Count of Participants; unit: Participants] — The HCT-CI is a comorbidity index that comprises 17 different categories of organ dysfunction. Positive findings are summated into a total score. The HCT-CI provides information with regard to the overall as well as non-relapse mortality risk a patient is likely to experience after hematopoietic cell transplantation. Lower scores have been shown to be associated with lower non relapse mortality.
  Participants
    0 | 9
    1 | 5
    2 | 15
    3 | 15
    4 | 10
    5 | 5
    6 | 8
    7 | 2
    8 | 1
    unknown | 2
Cytomegalovirus Status [Count of Participants; unit: Participants]
  CMV Seropositive | 45
  CMV Seronegative | 26
  unknown | 1
Disease [Count of Participants; unit: Participants]
  AML | 38
  ALL | 5
  MDS | 7
  Hodgkins | 3
  Non Hodgkins Lymphoma | 6
  Peripheral T cell Lymphoma | 3
  Other | 10
Remission Status [Count of Participants; unit: Participants]
  Complete Remission | 56
  Partial Remission | 9
  Stable Disease | 1
  Progressive Disease | 6
Minimal Residual Disease [Count of Participants; unit: Participants] — Population: Only patients in a complete remission were assessed for minimal residual disease. All others are known to have residual disease
  Participants
    number analyzed (Participants) | 56
    MRD positive | 36
    MRD negative | 19
    unknown | 1
Number of cord blood donors [Count of Participants; unit: Participants]
  Single Cord | 2
  Double Cord | 70
Level of HLA matching [Count of Participants; unit: Participants] — The standard for selecting unrelated umbilical cord blood units for transplantation for non-malignant diseases relies on antigen-level (lower resolution) HLA typing for HLA-A and HLA-B, and allele-level for HLA-DRB1. A 6 of 6 cord blood in matched at A, B and DR on both Haplotypes. 5 of 6 has one mismatch and 4 of 6 has 2 mismatched. 4 of 6 is commonly the maximum number of mismatches accepted for a cord blood transplant.
  Participants
    4/6 plus 4/6 | 27
    4/6 plus 5/6 | 19
    5/6 plus 5/6 | 19
    6/6 plus 6/6 | 4
    other | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Kaplan-Meier and cumulative incidence estimates will be used.
Time Frame: At 1 year
Measure: Number; unit: percent of patients
Groups:
- Treatment (Chemotherapy, Transplant): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6. Patients with low risk of graft failure (multi-agent chemotherapy in the last 3 months or history of autologous transplant) receive 200cGy TBI on day -1. Patients with high risk of graft failure receive 300 cGy TBI on day -1.
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.
  IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days 0 to +180 and mycophenolate mofetil IV or PO every 8 hours on days -3 to +96.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo umbilical cord blood transplant
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
percent of patients | 35

2. Secondary Outcome: Median Time to ANC > 500
Time Frame: By day 55
Measure: Median (Full Range); unit: days
Groups:
- Treatment (Chemotherapy, Transplant): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6. Patients with low risk of graft failure (multi-agent chemotherapy in the last 3 months or history of autologous transplant) receive 200cGy TBI on day -1. Patients with high risk of graft failure receive 300 cGy TBI on day -1.
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.
  IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days 0 to +180 and mycophenolate mofetil IV or PO every 8 hours on days -3 to +96.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo umbilical cord blood transplant
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV or PO
  Total-Body Irradiation: Undergo TBI
  Umbilical Cord Blood Transplantation: Undergo umbilical cord blood transplant
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
days | 18 [2 to 46]

3. Secondary Outcome: Number of Participants With Graft Failure/Rejection
Description: descriptive
Time Frame: By day 55
Measure: Number; unit: participants
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
participants | 3

4. Secondary Outcome: Time to Platelet Engraftment of > 20,000 Cells Per mm3
Description: median and range
Time Frame: By 6 months
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
days | 46 [7 to 161]

5. Secondary Outcome: Percent of Patients With Grade II-IV Acute Graft Versus Host Disease
Description: Chi-square test was used to determine percent of grade II-IV GVHD using Glucksberg criteria
Time Frame: By day 100
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
percent of patients | 67

6. Secondary Outcome: Percent of Patients With Acute GVHD Grades III-IV
Description: Fischer's exact test was used to determined percent of patients with acute grade III-IV GVHD by Glucksberg criteria
Time Frame: 100 days
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
percent of patients | 12

7. Secondary Outcome: Percent of Patients With Chronic GVHD
Description: Kaplan-Meier and cumulative incidence estimates will be used to measure percent of patients with chronic GVHD by NIH consensus criteria.
Time Frame: At 2 years
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
percent of patients | 19

8. Secondary Outcome: Percent of Patients With Non-relapse Mortality
Description: Kaplan-Meier and cumulative incidence estimates
Time Frame: 6 months
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
percent of patients | 21

9. Secondary Outcome: Percent of Patients With Non-relapse Mortality
Description: Kaplan-Meier and cumulative incidence estimates
Time Frame: 1 year
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 72
percent of patients | 38

ADVERSE EVENTS:
Time Frame: 100 days
Description: CTCAE Version 3.0
Groups:
- Treatment (Chemotherapy, Transplant): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 1-2 hours on day -6.
  Patients with low risk of graft failure receive 200 cGy TBI on day -1.
  Patients with high risk of graft failure receive 300 cGy TBI on day -1.
  UMBILICAL CORD BLOOD TRANSPLANT: Patients undergo donor umbilical cord blood infusion on day 0.
  IMMUNOSUPRESSIVE THERAPIES: Patients receive cyclosporine IV over 1 hour every 8-12 hours on days 0 to +180 and mycophenolate mofetil IV or PO every 8 hours on days -3 to +96.
Arm/Group | Treatment (Chemotherapy, Transplant)
All-Cause Mortality (participants affected / at risk) | 52/72
Serious Adverse Events (participants affected / at risk) | 18/72
Other Adverse Events (participants affected / at risk) | 59/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Transplant) (N=72)
Encephalopathy (Nervous system disorders) | 4 (4) — Likely related to a toxic or metabolic etiology
Syncope (Cardiac disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) — ARDS
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 2 (2)
Sepsis (Infections and infestations) | 3 (3)
Bladder Hemorrhage (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Intracerebral Hemorrhage (Nervous system disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Arrythmia (Cardiac disorders) | 1 (1) — atrial fibrillation and flutter
Fever and rash (Skin and subcutaneous tissue disorders) | 1 (1) — fever to 106 with generalized erythroderma
Encephalitis (Infections and infestations) | 1 (1) — HHV6
Hypertension (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Transplant) (N=72)
allergic reaction (Immune system disorders) | 2 (2)
hemolysis (Blood and lymphatic system disorders) | 1 (1)
orthostatic hypotension (Cardiac disorders) | 3 (3)
Thrombosis (Cardiac disorders) | 3 (3)
Left ventricular function decrease (Cardiac disorders) | 3 (3)
Troponin elevation (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 6 (6)
Arrythmia (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) — associated with GVHD
Hemolytic Anemia (Blood and lymphatic system disorders) | 1 (1)
Hemolytic Uremic syndrome (Renal and urinary disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 12 (12)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Infection-Lung (Infections and infestations) | 12 (12)
Infection-Blood (Infections and infestations) | 11 (22)
Infection-GU (Infections and infestations) | 12 (13)
Infection-GI (Infections and infestations) | 6 (6) — Includes stool
Infection-Oral Cavity (Infections and infestations) | 2 (3)
Febrile Neutropenia (Infections and infestations) | 25 (26)
Infection skin (Infections and infestations) | 2 (2)
Infection CNS (Infections and infestations) | 2 (2)
Infection-joint (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (17)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 4 (4)
Encephalopathy (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
Diffuse Alveolar Hemorrhage (Blood and lymphatic system disorders) | 6 (8)
Vaginal Bleeding (Renal and urinary disorders) | 1 (1)
Bladder Hemorrhage (Renal and urinary disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) — associated with GVHD
Mucositis (Gastrointestinal disorders) | 2 (2)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Patients were given 200 or 300 cGy TBI based on set definitions of high risk or low risk of graft failure. This was NOT a randomized study designed to show which dose of TBI was more effective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT00723099/Prot_SAP_000.pdf